CLINICAL TRIAL: NCT01152164
Title: Quality of Life in Patients After Combined Modality Treatment of Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Proff.assist. Vaneja Velenik, MD, PhD, Institute of Oncology
Other Study IDs: 125/08
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Rectal Cancer
Keywords: quality of life; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rectal cancer patients
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Quality of life assessment using questionnaires EORTC QLQ C30 and 38 at baseline, one year and two years after the surgery of rectal cancer, treated with preoperative capecitabine based radiochemotherapy
  Other Names: EORTC QLQ C30, EORTC QLQ C38

SUMMARY:
The goal of this study is gathering informations about patients' quality of life after combined modality treatment of rectal cancer to evaluate how combined modality treatment for rectal cancer affects patients' quality of life. The findings of this study may provide us important information that can be used in treatment decision and to develop programs to improve quality of life of patients with rectal cancer.

DETAILED DESCRIPTION:
Over the last two decades, rectal cancer research has lead to better understanding of disease behaviour, resulting in more efficient treatments and higher prevalence of cancer survivors.Due to aggressive therapy, rectal cancer survivors can exhibit late sequelae of treatment, most common being impaired bowel, voiding, sexual malfunctioning and quality of life impairment. In order to determine the impact of rectal cancer and its treatment on patients' quality of life over time, this study will prospectively follow a cohort of patients at specified intervals evaluating their physical symptoms, physical and social functioning and overall quality of life.Medical and sociodemographic factors that might be predictive will be tested.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified adenocarcinoma of the rectum,
* clinical stage II or III (IUCC TNM classification 2002);
* no prior radiotherapy and/or chemotherapy;
* World Health Organisation (WHO) performance status < 2;
* age at diagnosis of 18 or older;
* and adequate bone marrow, liver, renal and cardiac function (no history of ischemic heart disease)
* mentally fit to complete questionnaires

Exclusion Criteria:

* a history of prior malignancy other than non-melanoma skin cancer or in situ carcinoma of the cervix rendered the patient ineligible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with rectal cancer stage II and III, treated with capecitabine-based preoperative radiochemotherapy from 1.1.2008 till 31.12.2009.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2008-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate the quality of life of patients one year after rectal cancer resection | one year after the operation

SECONDARY OUTCOMES:
To prospectively evaluate the quality of life of patients at baseline | before treatment (at baseline)
  consecutive patients treated winh capecitabine-based radiochemotherapy
To prospectively evaluate the quality of life of patients two years after rectal cancer resection | two years after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia, Slovenia

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Sprangers MA, te Velde A, Aaronson NK. The construction and testing of the EORTC colorectal cancer-specific quality of life questionnaire module (QLQ-CR38). European Organization for Research and Treatment of Cancer Study Group on Quality of Life. Eur J Cancer. 1999 Feb;35(2):238-47. doi: 10.1016/s0959-8049(98)00357-8. PMID 10448266
- [Background] Moriya Y. Function preservation in rectal cancer surgery. Int J Clin Oncol. 2006 Oct;11(5):339-43. doi: 10.1007/s10147-006-0608-z. PMID 17058130
- [Background] Rauch P, Miny J, Conroy T, Neyton L, Guillemin F. Quality of life among disease-free survivors of rectal cancer. J Clin Oncol. 2004 Jan 15;22(2):354-60. doi: 10.1200/JCO.2004.03.137. PMID 14722043
- [Background] Parker PA, Baile WF, de Moor Cd, Cohen L. Psychosocial and demographic predictors of quality of life in a large sample of cancer patients. Psychooncology. 2003 Mar;12(2):183-93. doi: 10.1002/pon.635. PMID 12619150
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735